CLINICAL TRIAL: NCT05711628
Title: Randomized Phase III Trial of Chemotherapy vs. Pembrolizumab Plus Chemotherapy for Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: A Trial Comparing Chemotherapy Versus Novel Immune Checkpoint Inhibitor (Pembrolizumab) Plus Chemotherapy in Treating Relapsed/Refractory Classical Hodgkin Lymphoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Other - Protocol moved to Withdrawn
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-00575; NCI-2023-00575 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA4211 (Other: ECOG-ACRIN Cancer Research Group); EA4211 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-02-02; First posted 2023-02-03 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
MeSH Terms: interventions — Stem Cell Transplantation; Bendamustine Hydrochloride; Brentuximab Vedotin; Carboplatin; Etoposide; Gemcitabine; Ifosfamide; liposomal doxorubicin; Doxorubicin; pembrolizumab; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Transplantation Conditioning; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (chemotherapy regimen, HDT-ASCT) (Active Comparator): SALVAGE THERAPY: Patients receive 1 of 3 chemotherapy regimens as clinically indicated: 1) ifosfamide IV, carboplatin IV, and etoposide IV; 2) gemcitabine IV, vinorelbine IV, and pegylated liposomal doxorubicin IV; or 3) brentuximab vedotin IV and bendamustine IV. Patients then undergo a PET/CT scan. Patients who achieve a CR or PR proceed to HDT-ASCT. Patients who achieve SD or PD come off study treatment.
  HDT-ASCT: Patients undergo ASCT. Patients may also receive a standard preparative chemotherapy regimen as clinically indicated. Patients who achieve PR prior to ASCT may also undergo RT as clinically indicated. Patients who went into ASCT with PR also undergo a PET/CT scan 30 days post-transplant.
  MAINTENANCE THERAPY: Patients may receive brentuximab vedotin IV as clinically indicated.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Bendamustine; Drug: Brentuximab Vedotin; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Etoposide; Drug: Gemcitabine; Drug: Ifosfamide; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: Transplant Conditioning; Drug: Vinorelbine
- Arm B (chemotherapy regimens+pembrolizumab, HD-ASCT) (Experimental): SALVAGE THERAPY: Patients receive pembrolizumab IV plus 1 of 3 chemotherapy regimens specified in Arm A as clinically indicated. Patients then undergo a PET scan. Patients who achieve a CR or PR proceed to HDT-ASCT. Patients who achieve SD or PD come off study treatment.
  HDT-ASCT: Patients undergo ASCT. Patients may also receive a standard preparative chemotherapy regimen as clinically indicated. Patients who achieve PR prior to ASCT may also undergo RT as clinically indicated. Patients who went into ASCT with PR also undergo a PET/CT scan 30 days post-transplant.
  MAINTENANCE THERAPY: Patients may receive brentuximab vedotin IV as clinically indicated.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Bendamustine; Drug: Brentuximab Vedotin; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Etoposide; Drug: Gemcitabine; Drug: Ifosfamide; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: Transplant Conditioning; Drug: Vinorelbine

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Bendamustine — Given IV
  Other Names: SDX-105
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo PET/CT and CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475
  Arms: Arm B (chemotherapy regimens+pembrolizumab, HD-ASCT)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Other: Transplant Conditioning — Receive standard preparative chemotherapy regimen
  Other Names: conditioning regimen
Drug: Vinorelbine — Given IV
  Other Names: Dihydroxydeoxynorvinkaleukoblastine

SUMMARY:
This phase III trial compares chemotherapy versus an immune checkpoint inhibitor drug called pembrolizumab plus chemotherapy in treating patients with classical Hodgkin lymphoma that has come back (relapsed) or that does not respond to treatment (refractory). The usual approach for patients with classical Hodgkin lymphoma is treatment with standard chemotherapy, including drugs that are Food and Drug Administration (FDA)-approved. If this treatment puts a patient into remission, high dose chemotherapy and stem cell transplant may be used to increase the likelihood of a cure. Hodgkin lymphoma is capable of inhibiting the immune system from killing it. Pembrolizumab is a checkpoint inhibitor that may be able to stop this inhibition, allowing the immune system to attack the lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the 2-year event free survival (EFS) of patients treated with pembrolizumab added to chemotherapy versus chemotherapy alone, in patients with relapsed/refractory (R/R) classical Hodgkin's lymphoma (cHL) who are intended to receive salvage therapy followed by high dose chemotherapy and autologous stem cell transplant (HDT-ASCT).

PRIMARY IMAGING OBJECTIVE:

I. To assess the diagnostic performance of baseline total metabolic tumor volume (TMTV) in predicting response (complete remission [CR] + partial remission [PR] versus [vs] no response) at pre-transplant/post-salvage for each arm separately and overall.

SECONDARY OBJECTIVES:

I. To assess the 2-year progression free survival (PFS) and overall survival (OS) in the transplanted population.

II. To assess the complete remission (CR) rate to salvage therapy. III. To assess the CR rate post HDT-ASCT. IV. To assess the post HDT-ASCT partial remission (PR) to CR conversion rate.

SECONDARY IMAGING OBJECTIVES:

I. To assess the % change in TMTV (delta TMTV) from baseline to pre-transplant/post-salvage in predicting response (CR+PR vs no response) at pre-transplant/post-salvage for each arm separately and overall.

II. To assess baseline TMTV and delta TMTV in predicting EFS/OS for each arm separately and overall.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A:

SALVAGE THERAPY: Patients receive 1 of 3 chemotherapy regimens as clinically indicated: 1) ifosfamide intravenously (IV), carboplatin IV, and etoposide IV; 2) gemcitabine IV, vinorelbine IV, and pegylated liposomal doxorubicin IV; or 3) brentuximab vedotin IV and bendamustine IV. Patients then undergo a positron emission tomography (PET)/computed tomography (CT) scan. Patients who achieve a CR or PR proceed to HDT-ASCT. Patients who achieve stable disease (SD) or progressive disease (PD) come off study treatment.

HDT-ASCT: Patients undergo ASCT. Patients may also receive a standard preparative chemotherapy regimen as clinically indicated. Patients who achieve PR prior to ASCT may also undergo radiation therapy (RT) as clinically indicated. Patients who went into ASCT with PR also undergo a PET/CT scan 30 days post-transplant.

MAINTENANCE THERAPY: Patients may receive brentuximab vedotin IV as clinically indicated.

ARM B:

SALVAGE THERAPY: Patients receive pembrolizumab IV plus 1 of 3 chemotherapy regimens specified in Arm A as clinically indicated. Patients then undergo a PET scan. Patients who achieve a CR or PR proceed to HDT-ASCT. Patients who achieve SD or PD come off study treatment.

HDT-ASCT: Patients undergo ASCT. Patients may also receive a standard preparative chemotherapy regimen as clinically indicated. Patients who achieve PR prior to ASCT may also undergo RT as clinically indicated. Patients who went into ASCT with PR also undergo a PET/CT scan 30 days post-transplant.

MAINTENANCE THERAPY: Patients may receive brentuximab vedotin IV as clinically indicated.

All patients undergo CT scans during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 5 years of age and =< 75 years of age
* Patient must have relapsed/refractory classical Hodgkin lymphoma (R/R cHL) after frontline (first line of chemotherapy) as evidenced by Fludeoxyglucose F-18 (FDG) avid on PET scan. If regimen is adjusted based on PET2 results or toxicity during frontline therapy, this will only be considered one line of therapy. Prior checkpoint inhibitor is completed > 6 months prior to randomization
* Patients >= 18 years of age must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2. Pediatric patients (16-17 years of age) must have a Karnofsky performance level >= 50%. Pediatric patients (5-15 years of age) must have a Lansky performance level >= 50
* Patient must be deemed fit for high dose chemo and autologous stem cell transplant
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Pediatric patients (< 18 years of age) and patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible. Child assent must be obtained as appropriate in accordance with institutional guidelines
* Absolute neutrophil count (ANC) >= 1000/mcL (must be obtained =< 7 days prior to randomization)

  * If disease includes marrow involvement or hypersplenism, please reference the below revised requirement:

    * ANC >= 500/mcL
* Platelets >= 75,000/mcL (must be obtained =< 7 days prior to randomization)

  * If disease includes marrow involvement or hypersplenism, please reference the below revised requirement:

    * Platelets >= 25,000/mcL
* Total bilirubin =< 2x institutional upper limit of normal (ULN) (must be obtained =< 7 days prior to randomization)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN for age (must be obtained =< 7 days prior to randomization)
* Glomerular filtration rate (GFR) >= 50 mL/min/1.73m^2 73m^2 for patients >= 18 years of age (must be obtained =< 7 days prior to randomization)

  * Pediatric patients (< 18 years old) must have a creatinine clearance OR radioisotope GFR >= 70 mL/min/1.73 m^2 OR serum creatinine below the maximum based on age/gender as follows (derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention [CDC]):

    * Age: 5 to < 6 years; Maximum Serum Creatinine (mg/dL): Male (0.8); Female (0.8)
    * Age: 6 to 10 years; Maximum Serum Creatinine (mg/dL): Male (1.0); Female (1.0)
    * Age: 10 to 13 years; Maximum Serum Creatinine (mg/dL): Male (1.2); Female (1.2)
    * Age: 13 to < 16 years; Maximum Serum Creatinine (mg/dL): Male (1.5); Female (1.4)
    * Age: >= 16 years; Maximum Serum Creatinine (mg/dL): Male (1.7); Female (1.4)
* Patient must have a left ventricular ejection fraction (LVEF) >= 50%, as measured by echocardiogram, multi-gated acquisition (MUGA) scan, or functional cardiac imaging scan (or a shortening fraction of >= 27% for patients < 18 years of age only)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients >= 18 years of age with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better

Exclusion Criteria:

* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients of childbearing potential and/or sexually active patients must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study. Additionally, patients of childbearing potential must continue contraception measures for 4 months after the last dose of pembrolizumab, 6 months after the last dose of vinorelbine and for 3 months after the last dose of bendamustine. Male patients must continue contraception measures for 6 months after the last dose of ifosfamide and for 3 months after the last dose of vinorelbine. Patients must also not breastfeed while on study treatment and for 4 months after the last dose of Pembrolizumab and 9 days after the last dose of vinorelbine
* Patient must not have a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or have current pneumonitis/interstitial lung disease
* Patient must not have the following symptomatic autoimmune disorders: rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, Sjögren's syndrome, or autoimmune vasculitis (e.g., Wegener's Granulomatosis), or conditions of immunosuppression that require current ongoing treatment with systemic corticosteroids (or other systemic immunosuppressants), including oral steroids (i.e., prednisone, dexamethasone). Patients who discontinue use of these classes of medication for at least 2 weeks prior to randomization eligible if, in the judgment of the treating physician investigator, the patient is not likely to require resumption of treatment with these classes of drugs during the study.

  * Replacement doses of steroids for patients with adrenal insufficiency are allowed.
  * Additionally, patients must not have an autoimmune disease that is felt by the treating physician to have the potential to be exacerbated by checkpoint inhibition

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | Time from randomization to the earlier of events listed in description field, assessed up to 15 years
  Events include: failure to achieve partial remission (PR) or complete remission (CR) to salvage chemotherapy, failure to achieve a CR post high dose chemotherapy and autologous stem cell transplant (HDT-ASCT), progression, receipt of unplanned radiation or brentuximab vedotin maintenance, or death. Patients who have not experienced any of these events will be censored at the date they are last known to be progression free. Kaplan-Meier method will be used to estimate EFS, including medians and confidence intervals. Comparison of EFS between treatment arms will be conducted based on intent-to-treat principle using a one-sided stratified log-rank test with the stratification factors.
Lugano-based response | Pre-transplant/post-salvage therapy
  Will be assessed using positron emission tomography/computed tomography (PET/CT) scan with Deauville score. Will assess the diagnostic performance of baseline metabolic tumor volume (TMTV) in predicting response (CR+PR vs no response) at pre-transplant/post-salvage, overall and by study arm. Diagnostic performance of baseline TMTV will be assessed using area under the receiver operator characteristic curve (ROC AUC) analysis, where the reference standard is pre-transplant/post-salvage response (CR/PR).

SECONDARY OUTCOMES:
Percentage change in TMTV (delta TMTV) | Baseline to pre-transplant/post-salvage therapy
  Similar methods will be used as the primary imaging aim to assess the diagnostic performance of delta TMTV in predicting pre-transplant/post-salvage response (CR+PR vs no response). Delta TMTV will be defined as the percent change from baseline to pre-transplant/post-salvage [(post-salvage/pre-transplant - baseline)/baseline X 100].
Baseline TMTV and delta TMTV | Baseline and pre-transplant/post-salvage therapy
  Will assess baseline TMTV and delta TMTV in predicting EFS/overall survival (OS) for each arm separately and overall. The association between TMTV and EFS will be analyzed through a Cox regression model. TMTV will be analyzed individually as its absolute value and the percent change from baseline. We will also test if there is a difference by arm by including an interaction term in the model between TMTV and arm. The Kaplan-Meier method will be used to estimate EFS, including median survival times and confidence intervals. In addition to examining the TMTV, we will also analyze standard uptake value maximum (SUVmax) and total lesion glycolysis (TLG) with the same methods. The OS outcome will be analyzed in a similar manner.

CONTACTS AND LOCATIONS:
Overall Officials: Vaishalee P Kenkre, Principal Investigator — ECOG-ACRIN Cancer Research Group

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm